CLINICAL TRIAL: NCT00137852
Title: Phase II Trial of Cisplatin, CPT-11, Celecoxib (PCC), Concurrent Radiation Therapy, and Surgery for Resectable Esophageal Cancer
Brief Title: Cisplatin, CPT-11 and Celecoxib With Radiation Therapy and Surgery for Operable Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Pharmacia (Industry)
Responsible Party: Principal Investigator, Peter C. Enzinger, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-229
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Esophageal Cancer
Keywords: Esophageal Cancer; Resectable Esophageal Cancer; Radiation Therapy; Celecoxib; Irinotecan; Cisplatin
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Cisplatin; Irinotecan; Celecoxib; Radiotherapy; Esophagectomy

ARMS (1):
- Cisplatin/CPT-11/Celecoxib/XRT/Surgery (Experimental): Cisplatin, CPT-11 and Celecoxib With Radiation Therapy and Surgery for Operable Esophageal Cancer
  Interventions: Drug: Cisplatin; Drug: Irinotecan; Drug: Celecoxib; Procedure: Radiation Therapy; Procedure: Esophagectomy

INTERVENTIONS:
Drug: Cisplatin — Given weekly on weeks 1, 2, 4 and 5 during radiation therapy.
Drug: Irinotecan — Given weekly on weeks 1, 2, 4 and 5 during radiation therapy
  Other Names: CPT-11
Drug: Celecoxib — Given twice daily 3 days prior to radiation and up until one week prior to surgery. It will then be started again once the participant is released from the hospital following surgery for 26 weeks.
Procedure: Radiation Therapy — 5 days a week for 5-6 weeks
Procedure: Esophagectomy — Within 4-8 weeks of chemoradiation therapy

SUMMARY:
This is a study for patients with resectable, locally advanced esophageal cancer. There is evidence to suggest that celecoxib in combination with cisplatin and irinotecan (CPT-11) may work well with radiation therapy to kill cancer cells. The primary goal is to develop a well-tolerated cancer treatment that has an acceptable response rate.

DETAILED DESCRIPTION:
Patients will take celecoxib orally twice daily 3 days prior to radiation therapy and until one week prior to surgery. Celecoxib will then be restarted when the patient is discharged from the hospital following surgery and continued for 26 weeks.

Patients will receive chemotherapy (cisplatin and irinotecan) weekly on weeks 1, 2, 4 and 5 during radiation therapy. Chemotherapy must occur on or before the fifth day of radiation therapy.

Radiation therapy will be performed 5 days a week over a 5.6 week period.

Patients will undergo an esophagectomy within 4-8 weeks of chemotherapy/radiation therapy. Technically accessible lymph nodes will also be removed.

During chemotherapy/radiation therapy, a physical exam and bloodwork will be conducted weekly.

Between chemotherapy/radiation therapy and surgery a physical exam, bloodwork and CT of chest, abdomen, and pelvis should be performed.

After the completion of treatment and surgery, a physical exam and bloodwork should be done every 6 weeks for 6 months, then every 3 months for 1 1/2 years, then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years.
* Adenocarcinoma or squamous cell carcinoma of the esophagus, including the gastroesophageal junction, histologically confirmed, American Joint Committee on Cancer (AJCC) Stage IIA, IIB, III. Additionally, patients with tumors of the lower thoracic esophagus and gastroesophageal junction may have regional lymph node involvement (M1A-Stage IVA), as long as the lymphadenopathy can be entirely encompassed by the radiation field.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Neutrophils greater than or equal to 1,500/ μL.
* Platelets greater than or equal to 100,000/ μL.
* Serum bilirubin less than or equal to 1.5 mg/dl.
* Serum creatinine less than or equal to 1.5 mg/dl.
* Aspartamine transaminase (AST or SGOT) less than or equal to 3x upper institutional normal limit.
* Alkaline phosphatase less than or equal to 5x upper institutional normal limit.

Exclusion Criteria:

* No prior surgery for esophageal or gastro-esophageal junction cancer.
* No prior chemotherapy or radiation therapy.
* Biopsy proven tumor invasion of the tracheobronchial tree or a tracheoesophageal fistula.
* Metastatic disease to distant organs (e.g. liver, lungs, bone) or non-regional lymph nodes. Patients with supraclavicular/cervical lymph node involvement or patients with a proximal esophageal primary and celiac/gastro-hepatic lymph node involvement are also excluded.
* Patients with co-morbid disease that, in the opinion of the investigator, makes combined chemo-radiotherapy inadvisable (e.g. New York State Grade III-IV heart disease, myocardial infarction in the last 4 months, uncontrolled infection, uncontrolled diabetes, uncontrolled hypertension, uncontrolled psychiatric illness or organ allograft(s) on immunosuppressive therapy).
* Pregnant or lactating women or women of childbearing potential with either a positive or no pregnancy test at baseline.
* Women of childbearing potential not using a reliable and appropriate contraceptive method. (Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential.)
* Other active malignancy (i.e. hematologic malignancy, metastatic solid tumor, or resected Stage I-IV solid tumor less than 3 years after resection).
* Patients with known Gilbert's disease or interstitial pulmonary fibrosis.
* Patients with prior severe reaction to nonsteroidal anti-inflammatory drugs (NSAIDs), sulfonamides, or celecoxib.
* Patients with a history of seizure disorders who are receiving antiepileptic medication.
* Positive malignant cytology of the pleura, pericardium or peritoneum.
* Uncontrolled diarrhea (National Cancer Institute Common Toxicity Criteria [NCI CTC] greater than or equal to Grade 2).
* Peripheral neuropathy (NCI CTC greater than or equal to Grade 2).
* Symptomatic hearing loss, requiring a hearing aid or for which a hearing aid has been suggested by a health professional.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2002-01; Primary Completion 2004-08 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Response rate of combination of chemotherapy, radiation therapy and surgery in resectable esophageal carcinoma

SECONDARY OUTCOMES:
Determine the side effects of chemotherapy and radiation therapy in patients with resectable esophageal carcinoma | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter C. Enzinger, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Result] Cleary JM, Mamon HJ, Szymonifka J, Bueno R, Choi N, Donahue DM, Fidias PM, Gaissert HA, Jaklitsch MT, Kulke MH, Lynch TP, Mentzer SJ, Meyerhardt JA, Swanson RS, Wain J, Fuchs CS, Enzinger PC. Neoadjuvant irinotecan, cisplatin, and concurrent radiation therapy with celecoxib for patients with locally advanced esophageal cancer. BMC Cancer. 2016 Jul 13;16:468. doi: 10.1186/s12885-016-2485-9. PMID 27412386